CLINICAL TRIAL: NCT05912647
Title: A Multiphase Optimization Strategy to Enhance Diabetes Management Interventions for Patients With Uncontrolled Diabetes
Brief Title: Enhancing Diabetes Management Approaches for Patients With Uncontrolled Diabetes
Acronym: ENRxICH
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Wisconsin, Madison (Other)
Collaborators: National Institute of Diabetes and Digestive and Kidney Diseases (NIDDK) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: 2023-0780; 1R01DK136690-01 (NIH); PHARM/PHARMACY (Other: UW Madison); Protocol Version 5/23/25 (Other: UW Madison)
Record Dates: First submitted 2023-06-12; First posted 2023-06-22 (Actual); Last update posted 2025-08-14 (Actual); Status verified 2025-08

CONDITIONS: Diabetes; Diabetes Type 2
MeSH Terms: conditions — Diabetes Mellitus; Diabetes Mellitus, Type 2

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (4):
- Usual Care (No Intervention)
- Medication Therapy Management (MTM) (Experimental)
  Interventions: Behavioral: MTM
- Community Health Worker (CHW) (Experimental)
  Interventions: Behavioral: CHW
- MTM + CHW (Experimental)
  Interventions: Behavioral: MTM; Behavioral: CHW

INTERVENTIONS:
Behavioral: MTM — Participants will receive added medicine management support from a pharmacist. This will involve one 60-minute session with the pharmacist either in-person or over the phone and at least four 30-minute follow-up sessions with the pharmacist over the phone.
  Arms: MTM + CHW; Medication Therapy Management (MTM)
Behavioral: CHW — Participants will receive support from a Community Health Worker (CHW) to address life challenges that might be affecting their health and diabetes and to discuss diabetes beliefs and concerns. This will involve one ~30-minute phone call with the CHW to discuss needs and a 2-hour session with the CHW in-person for a comprehensive assessment. Participants will also receive ~10, 15 to 30-minute calls from the CHW to discuss diabetes beliefs and concerns.
  Arms: Community Health Worker (CHW); MTM + CHW

SUMMARY:
The purpose of the study is to learn about the best way to enhance pharmacy-related care for diabetes self-management.

This research is being done because we want to improve use of medicines and diabetes management among adults with type 2 diabetes and find out which of type of support may improve diabetes self-management for adults.

Participants will be assigned to one of 4 groups, and will either:

* receive care as usual; or,
* receive added medicine management support from a pharmacist; or,
* receive support from a Community Health Worker (CHW) to address life challenges; or,
* receive both the pharmacist medicine management and the CHW support

DETAILED DESCRIPTION:
For the ENRxICH intervention, all participants will receive usual care for their diabetes management. Participants will be randomized to one of four treatment conditions: 1. Usual Care, 2. Medication Therapy Management (MTM) Optimizing Medication Therapy (ON), 3. Community Health Worker (CHW) addressing social determinants of health (SDOH) and diabetes and medicine misperceptions (ON), or 4. both MTM Optimizing Medication Therapy and CHW Addressing SDOH and diabetes and medicine misperceptions for 6 months.

Subjects randomized to the treatment conditions including MTM will receive a minimum of five pharmacist-delivered Medication Therapy Management (MTM) sessions with a pharmacist, two in the first month, one medication review each in the second and third month, and a final medication review at 6 months.

Subjects randomized to the treatment conditions including CHW support addressing social determinants of health (SDOH) which will involve meeting with the CHW for a formal, standardized 2-hour assessment of five common SDOH barriers related to diabetes management, (1) food insecurity, (2) transportation, (3) prescription medication assistance, (4) access to diabetes education, and (5) physical activity resources (See Table 6). After the initial session at the participant's home (or another community location), the participant will have the option of continuing to work with the CHW to address barriers for the intervention duration. CHW support will also address diabetes and medicine misperceptions by completing a series of phone calls with the subject to provide information about managing diabetes and medicines, discuss cultural health misperceptions, share medication adherence experiences, and provide social support over the phone.

ELIGIBILITY:
Inclusion Criteria:

* Men and women ages 18-90 with diagnosed type 2 diabetes who speak and understand English or Spanish.
* Taking at least one oral or injectable diabetes medication
* HbA1c ≥ 8% based on point of care test.
* Will reside in the geographical area throughout the study period.
* Have access to a phone during the study period.
* Willing to attend all orientation/training sessions.

Exclusion Criteria:

* Having a caregiver who is the main decision maker in self-management.
* Participating in another lifestyle, or medication adherence program.
* Participated in standard MTM/MTM-related intervention in the last 6 months.

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 376 (Estimated)
Dates: Start 2024-02-03 (Actual); Primary Completion 2027-12 (Estimated); Study Completion 2027-12 (Estimated)

PRIMARY OUTCOMES:
Change in mean hemoglobin A1c score | Baseline to 6 months
  HbA1c will be measured, and the mean change will be compared across arms
Change in mean hemoglobin A1c score | Baseline to 12 months
  HbA1c will be measured, and the mean change will be compared across arms

SECONDARY OUTCOMES:
Change in medication adherence - medication refill | 6 months and 12 months
  Pharmacy medication refill measured by Proportion of Days Covered and Medication Possession Ratio in subjects receiving MTM, CHW support, or both, compared to those receiving usual care.
Mean scores on the Adherence to Refills and Medications Scale for Diabetes | 6 months and 12 months
  Mean scores on the Adherence to Refills and Medications Scale for Diabetes in subjects receiving MTM, CHW support, or both, compared to those receiving usual care. The scores range from 11-44, lower scores indicate better medication adherence.

CONTACTS AND LOCATIONS:
Overall Officials: Michelle Chui, PharmD, PhD, Principal Investigator — University of Wisconsin, Madison
Locations (1):
- University of Wisconsin, Madison, Wisconsin, United States

IPD SHARING:
Plan to Share IPD: Yes
Supporting Information: Study Protocol, SAP, ICF